CLINICAL TRIAL: NCT04420884
Title: An Open-label, Dose Escalation, Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAK-676 as a Single Agent and in Combination With Pembrolizumab in Adult Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of Dazostinag as Single Agent and Dazostinag in Combination With Pembrolizumab in Adults With Advanced or Metastatic Solid Tumors
Acronym: iintune-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-676-1002; U1111-1241-4427 (Registry Identifier: WHO); 2023-505627-30-00 (EU CTIS Number: EU CT Number); jRCT2031230532 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Solid Neoplasms
Keywords: Drug Therapy
MeSH Terms: interventions — pembrolizumab; Platinum; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1 (Monotherapy Dose Escalation Phase): Dazostinag Safety Lead-in + Dazostinag SA [Part 1A] (Experimental): Safety Lead-in: Dazostinag 0.1 mg, infusion, intravenously (IV), once weekly, on Days 1, 8 and 15 in 21-day treatment cycles.
  Dazostinag SA Dose Escalation (Part 1A): Dazostinag single agent (SA), infusion, IV, once weekly on Days 1, 8 and 15 in each 21-day treatment cycles with escalating doses (0.2 mg and above). The dosing will be initiated in the Dazostinag SA Dose Escalation Phase based on the available safety and tolerability data from the Safety Lead-in.
  Interventions: Drug: Dazostinag
- Part 1B (Combination Dose Escalation Phase): Dazostinag + Pembrolizumab (Experimental): Dazostinag escalating doses (0.2 mg and above) in combination with pembrolizumab 200 mg, infusion, IV, once weekly on Days 1, 8 and 15 in each 21-day treatment cycle. Pembrolizumab 200 mg will be administered 1 hour prior to Dazostinag once every 3 weeks (Q3W). The dosing will be initiated when at least two dose levels (DLs) of Part 1A have been evaluated.
  Interventions: Drug: Dazostinag; Drug: Pembrolizumab
- Arm A: Japan Safety Lead-in Dazostinag + Pembrolizumab (Experimental): Dazostinag 5.0 mg, infusion, IV, in Japanese participants with advanced or metastatic solid tumors on Days 1, 8, and 15 in each 21-day cycle in combination with pembrolizumab 200 mg administered Q3W, IV, on Day 1 in each 21-day cycle.
  Additional dose levels of Dazostinag (such as 14.0 mg) in combination with pembrolizumab (200 mg, Q3W) may be explored in the Safety Lead-in.
  Interventions: Drug: Dazostinag; Drug: Pembrolizumab
- Arm B: Japan Safety Lead-in Dazostinag Transitioned to Pembrolizumab (Experimental): Dazostinag 5.0 mg, infusion, IV, as an SA once on Day 1 in Cycle 0 (cycle length=7 days) in Japanese participants with advanced or metastatic solid tumors based on confirmation of tolerability in Arm A. Following Cycle 0 (7 days), participants will be transitioned to the same dose level of dazostinag on Days 1, 8, and 15 of each 21-day cycle in combination with pembrolizumab administered Q3W, IV, on Day 1 in each 21-day cycle.
  Additional dose levels of dazostinag (such as ≥ 7.0 mg) in combination with pembrolizumab (200 mg, Q3W) may be explored in the Safety Lead-in.
  Interventions: Drug: Dazostinag; Drug: Pembrolizumab
- Part 2A (SCCHN CPS ≥ 1 Dose Expansion and Optimization Phase): Dazostinag + Pembrolizumab (Experimental): Dazostinag 5.0 mg, infusion, IV, will be administered in participants with squamous cell carcinoma of head and neck (SCCHN) at the identified dose level from Part 1 on Days 1, 8, and 15 in a 21-day cycle along with pembrolizumab 200 mg infusion, IV, Q3W. Dose optimization may be performed in this phase.
  Interventions: Drug: Dazostinag; Drug: Pembrolizumab
- Part 2B (SCCHN Dose Expansion Phase): Dazostinag + Pembrolizumab + Chemotherapy (Experimental): Dazostinag 5.0 mg, infusion, IV, will be administered in participants with SCCHN at the identified dose level from Part 1 on Days 1, 8, and 15 in a 21-day cycle. Pembrolizumab infusion, IV will be administered at 200 mg Q3W. Platinum-based chemotherapy comprising the combination of carboplatin (target area under the curve of 5 milligrams per milli Liters per minute (mg/mL/minute) [AUC 5]) or cisplatin (100 milligrams per square meter [mg/m^2] Day 1 of each treatment cycle), and 5-fluorouracil ([5-FU]; 1000 mg/m^2 per day for 4 consecutive days) Q3W for up to 6 cycles.
  Interventions: Drug: Dazostinag; Drug: Pembrolizumab; Drug: Platinum; Drug: 5-fluorouracil
- Part 3A (Expansion Phase in CRC): Dazostinag + Pembrolizumab in MSI-H/dMMR CRC (Experimental): Dazostinag 5.0 mg, infusion, IV, will be administered in participants with microsatellite instability-high /mismatch repair deficient (MSI-H/dMMR) colorectal cancer (CRC) at the identified dose level from Part 1 on Days 1, 8, and 15 in a 21-day cycle along with pembrolizumab 200 mg infusion, IV, Q3W.
  Interventions: Drug: Dazostinag; Drug: Pembrolizumab
- Part 3B (Expansion Phase in CRC): Dazostinag + Pembrolizumab in MSS/pMMR CRC (Experimental): Dazostinag 5.0 mg, infusion, IV, will be administered in participants with microsatellite stable/mismatch repair proficient (MSS/pMMR) CRC at the identified dose level from Part 1 on Days 1, 8, and 15 in a 21-day cycle. along with pembrolizumab 200 mg infusion, IV, Q3W.
  Interventions: Drug: Dazostinag; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Dazostinag — Dazostinag intravenous infusion.
  Other Names: TAK-676
Drug: Pembrolizumab — Pembrolizumab intravenous infusion.
  Arms: Arm A: Japan Safety Lead-in Dazostinag + Pembrolizumab; Arm B: Japan Safety Lead-in Dazostinag Transitioned to Pembrolizumab; Part 1B (Combination Dose Escalation Phase): Dazostinag + Pembrolizumab; Part 2A (SCCHN CPS ≥ 1 Dose Expansion and Optimization Phase): Dazostinag + Pembrolizumab; Part 2B (SCCHN Dose Expansion Phase): Dazostinag + Pembrolizumab + Chemotherapy; Part 3A (Expansion Phase in CRC): Dazostinag + Pembrolizumab in MSI-H/dMMR CRC; Part 3B (Expansion Phase in CRC): Dazostinag + Pembrolizumab in MSS/pMMR CRC
Drug: Platinum — Carboplatin or Cisplatin intravenous infusion
  Arms: Part 2B (SCCHN Dose Expansion Phase): Dazostinag + Pembrolizumab + Chemotherapy
Drug: 5-fluorouracil — 5-fluorouracil intravenous infusion
  Arms: Part 2B (SCCHN Dose Expansion Phase): Dazostinag + Pembrolizumab + Chemotherapy

SUMMARY:
The main aim of this study is to check if people with advanced solid tumors have side effects from dazostinag, and to check how much dazostinag they can receive without getting significant side effects from it when given alone and in combination with pembrolizumab. The study will be conducted in two phases including a dose escalation phase and a dose expansion phase. In the dose escalation phase, escalating doses of dazostinag are being tested alone and in combination with pembrolizumab to treat participants who have advanced or metastatic solid tumors. In the dose expansion phase, dazostinag will be studied with pembrolizumab with or without chemotherapy in participants with untreated metastatic or recurrent, unresectable squamous cell carcinoma of head and neck (SCCHN) and in combination with pembrolizumab in third-line or later recurrent locally advanced or metastatic microsatellite instability-high/mismatch repair deficient (MSI-H/dMMR) and third-line recurrent locally advanced or metastatic microsatellite stable/mismatch repair proficient (MSS/pMMR) colorectal cancer (CRC).

DETAILED DESCRIPTION:
The drug being tested in this study is called dazostinag. Dazostinag is being tested to treat people who have advanced or metastatic solid tumors.

The study will enroll approximately 374 participants. Part 1 consists of an initial Safety Lead-in to Dose Escalation Phase; Part 2 and Part 3 compose the Expansion Phase in 2 specific indications namely, previously untreated metastatic or recurrent, unresectable SCCHN (Part 2) and third-line or later recurrent locally advanced or metastatic MSI-H/dMMR and third-line recurrent locally advanced or metastatic MSS/pMMR CRC (Part 3). Participants will be assigned to the following treatment groups in the respective Phases of the study:

* Part 1 (Dose Escalation Phase): Safety Lead-in + Dazostinag single agent (SA) [Part 1A] Dazostinag 0.1 milligram (mg) in the Safety Lead-in followed by Dazostinag as escalating doses (0.2 mg and above) in Part 1A
* Part 1B (Combination Dose Escalation Phase): Dazostinag as escalating doses (0.2 mg and above) + Pembrolizumab
* Japan Safety Lead-in: Dazostinag SA 5.0 mg in the Safety Lead-in± Pembrolizumab in Arms A and B. Additional dose levels of Dazostinag (such as 14.0 mg) in combination with pembrolizumab may be explored during the Japan safety lead-in considering recommended dose for expansion (RDE1) as 5.0 mg and dose optimization.

Once a safe dose is recommended from Part 1, participants of select advanced or metastatic solid tumors will receive dazostinag in below defined cohorts in the expansion phase:

* Part 2A (SCCHN Combined Positive Score [CPS] ≥ 1 Dose Expansion Phase): Dazostinag + Pembrolizumab*
* Part 2B (SCCHN Dose Expansion Phase): Dazostinag + Pembrolizumab + Chemotherapy
* Part 3A (Expansion Phase in CRC): Dazostinag + Pembrolizumab in MSI-H/dMMR CRC
* Part 3B (Expansion Phase in CRC): Dazostinag + Pembrolizumab in MSS/pMMR CRC

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 68 months. Participants will make multiple visits to the clinic, including 30 days after last dose of study drug for a follow-up assessment. Participants in Parts 2 and 3 will be followed for survival for up to 12 months after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
2. Dazostinag SA (dose escalation Part 1A):

   o With histologically confirmed (cytological diagnosis is acceptable) advanced or metastatic solid tumors that have no standard therapeutic options or are intolerant to these therapies.
3. Dazostinag in combination with pembrolizumab (dose escalation Parts 1B and Japan safety lead-in):

   * With histologically confirmed (cytological diagnosis is acceptable) advanced or metastatic solid tumors that have no standard therapeutic options or are intolerant to them, including:
   * Tumors that have relapsed or are refractory to anti-programmed cell death ligand protein 1 (anti PD-(L)-1) therapy.
   * Tumors that are naive to anti-PD-(L)-1 therapy.
4. For expansion phase only:

   * SCCHN (Part 2):
   * Participants with histologically confirmed (cytological diagnosis is acceptable) metastatic or recurrent, unresectable SCCHN that is considered incurable by local therapies. Participants should not have had prior systemic therapy administered in the recurrent or metastatic setting. Systemic therapy which was completed more than 6 months before signing consent if given as part of multimodal treatment of locally advanced disease is allowed.
   * Anatomic subsites to be included are oral cavity, oropharynx, hypopharynx, larynx, nasal cavity, and paranasal sinuses (maxillary, ethmoid, sphenoid, and frontal). The exception to this is nasopharyngeal cancer and salivary gland tumors, which will not be included.
   * Participants with oropharyngeal cancer or tumors arising in the paranasal sinuses (maxillary, ethmoid, sphenoid, and frontal) must agree to provide archival tissue for human papilloma virus (HPV) testing or if known, HPV testing results (using CINtec® p16 Histology assay is preferred but not required) and a 70% cutoff point must be provided. Alternatively, archival tissue or a fresh excisional or core needle biopsy (≥ 2 cores) is required for the determination of HPV status. If HPV status was previously tested using this method (CINtec® p16 Histology assay is preferred but not required), no additional testing is required. Archival tissue can be obtained up to 90 days prior to screening. Samples that are older than 90 days at screening may be used after consultation with the sponsor.
   * For Part 2A, tumors must have a PD-L1 CPS ≥ 1. Participants must agree to provide fresh tumor biopsy for analysis from a core or excisional biopsy (fine needle aspirate is not sufficient) at screening for PD-L1 CPS assessment by a central laboratory. This specimen may be the diagnostic sample for participants with a new diagnosis of metastatic SCCHN. Participants for whom newly obtained samples cannot be obtained (eg, inaccessible or participant safety concern) may submit an archived specimen only upon agreement from the Sponsor. Archival tissue can be obtained up to 90 days prior to screening provided there was no other treatment from the time of biopsy until the start of study treatment. For Part 2B, any CPS is eligible but fresh or archival tissue is required for confirmation of CPS status. Collection of the tissue samples for PD-L1 assessments for Part 2B can be discontinued by the sponsor if sufficient data has been collected or dazostinag activity does not justify further collection.
   * For Part 2B, participants must be eligible to receive treatment with either cisplatin or carboplatin in combination with 5-fluorouracil (5-FU) per the treating physician.
5. CRC (Part 3):

   * Third-line or later MSI-H/dMMR CRC (Part 3A): Participants with histologically confirmed (cytological diagnosis is acceptable) recurrent locally advanced or metastatic MSI-H/dMMR CRC whose disease has progressed on or following therapy with 1) an anti-PD-1 or PD-L1 antibody (i.e., pembrolizumab) and 2) at least one line of combination chemotherapy including a fluoropyrimidine and irinotecan OR oxaliplatin with or without an anti-epidermal growth factor receptor (EGFR) or anti-vascular endothelial growth factor (VEGFR) monoclonal antibody (i.e., cetuximab or bevacizumab). MSI-H/dMMR CRC participants must have received at least 6 weeks of prior treatment with an anti-PD-(L)-1 antibody. Only one line of anti-PD-(L)-1 is permitted.
   * Third-line MSS/pMMR CRC (Part 3B): Participants with histologically confirmed (cytological diagnosis is acceptable) recurrent locally advanced or metastatic MSS/pMMR CRC whose disease has progressed on or following therapy with 2 different lines of combination chemotherapy, including therapy with a fluoropyrimidine and irinotecan AND therapy with a fluoropyrimidine and oxaliplatin. Both lines of therapy may be given with or without an anti-EGFR or anti-VEGFR monoclonal antibody (i.e., cetuximab or bevacizumab).

   Participants with MSS/pMMR CRC must have progressed on or after combination chemotherapy regimens containing BOTH irinotecan AND oxaliplatin.
   * Participants with MSI-H/dMMR or MSS/pMMR CRC must have documented MSI/MMR status assessed by a Clinical Laboratory Improvements Amendment-certified (United States [US] sites or an accredited (outside of the US) local laboratory using immunohistochemistry (IHC) and/or polymerase chain reaction (PCR) or next generation sequencing (NGS) assay.
   * Adequate tumor tissue available for central laboratory confirmation of MSI/MMR status. Note: confirmation of central test positivity is not required before treatment.
   * Participants with MSI-H/dMMR or MSS/pMMR CRC must have been treated with 2 prior lines of therapy in the recurrent locally advanced or metastatic setting.
6. Adequate bone marrow, renal, hepatic and cardiac functions.
7. Left ventricular ejection fraction (LVEF) > 50%, as measured by echocardiogram or multiple-gated acquisition (MUGA) scan within 4 weeks before receiving the first dose of study drug.
8. Clinically significant toxic effects of previous therapy have recovered to Grade 1 (per NCI CTCAE Version 5.0) or baseline, except for alopecia, Grade 2 peripheral neuropathy, and/or autoimmune endocrinopathies with stable endocrine replacement therapy.
9. In dose escalation Part 1, (not applicable for the Japan safety lead-in) once peripheral evidence of dazostinag pharmacodynamic stimulation of the innate and/or adaptive immune system is observed in the blood and/or an imaging response/partial response (CR/PR) is observed in at least 1 participant, subsequent participants must:

   * Have at least 1 lesion amenable for biopsy.
   * Agree to have 2 tumor biopsies: 1 during the screening period and 1 while on dazostinag treatment.
10. Must have at least 1 RECIST version 1.1-evaluable (measurable) lesion. For the dose escalation phase (Part 1) only, nonmeasurable only disease is acceptable.
11. Pharmacokinetic (PK)/pharmacodynamic blood must be drawn on a peripherally-inserted catheter. Dazostinag is preferentially administered through a central line, but peripheral infusion is acceptable. If a peripheral line is used for dazostinag and/or pembrolizumab infusion, it must be separate than the one used for PK/pharmacodynamic collection.

Exclusion Criteria:

1. Corrected QT interval by Fredericia (QTcF) greater than (>) 450 milliseconds (men) or > 475 milliseconds (women) on a 12-lead electrocardiogram (ECG) during the screening period.
2. Grade greater than or equal to (≥) 2 hypotension (that is, hypotension for which nonurgent intervention is required) at screening or during Cycle 0 Day 1 (C0D1) [for Japan safety lead-in only] and Cycle 1 Day 1 (C1D1) predose assessment.
3. Oxygen saturation less than (<) 92 percent (%) on room air at screening or during C0D1 (for Japan safety lead-in only) and C1D1 predose assessment.
4. Treated with other STING agonists/antagonist and toll-like receptors agonists within the past 6 months.
5. Current history of pneumonitis, interstitial lung disease, severe chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, other restrictive lung diseases, acute pulmonary embolism, or Grade ≥ 2 pleural effusion or ascites not controlled by tap or requiring indwelling catheters.
6. History of brain and leptomeningeal metastasis unless:

   * Brain metastases are clinically and radiologically stable or improved (that is, ≥ 4 weeks) following surgery, whole-brain radiation, or stereotactic radiosurgery, AND
   * Off corticosteroids.
7. Ongoing Grade ≥ 2 infection or participants with Grade ≥ 2 fever of malignant origin.
8. Chronic, active hepatitis (example: participants with known hepatitis B surface antigen seropositive and/or detectable hepatitis C virus [HCV]- ribonucleic acid [RNA]).
9. For participants in the dose escalation SA Part 1A only: refusal of standard therapeutic options.
10. For participants receiving pembrolizumab only: contraindication and/or intolerance to the administration of pembrolizumab.
11. For participants receiving chemotherapy in Part 2B: contraindication and/or intolerance to the administration of both platinum agents (cisplatin and carboplatin) and/or 5-FU.
12. Participant has had any other prior or concurrent malignancy within 2 years prior to enrollment with the following exceptions: adequately treated localized basal cell or squamous cell carcinoma, or curatively treated in situ carcinoma of the cervix or breast. Other exceptions may be considered upon sponsor consultation.
13. Concurrent chemotherapy (except for Part 2B), immunotherapy (except for pembrolizumab in Part 1B, Part 2, and Part 3), biologic, or hormonal therapy (except for adjuvant endocrine therapy for a history of breast cancer). Concurrent use of hormones for noncancer-related conditions is acceptable (except for corticosteroid hormones) unless allowed per exclusion criterion 16.
14. Radiation therapy within 14 days (42 days for radiation to the lungs) and/or systemic treatment with radionuclides within 42 days before C1D1 of study drug(s). Participants with clinically relevant ongoing pulmonary complications from prior radiation therapy are not eligible.
15. Use of systemic corticosteroids or other immunosuppressive therapy, concurrently or within 7 days of C1D1 of study drug(s), with the following exceptions:

    * Topical, intranasal, inhaled, ocular, intra-articular, and/or other non-systemic corticosteroids.
    * Premedications required for computed tomography (CT) or magnetic resonance imaging (MRI) scans.
    * Physiological doses of replacement steroid therapy (example: for adrenal insufficiency).
    * For participants enrolled in Part 2B, chemotherapy premedication with steroids can be administered according to local standards of care practice.
16. Use of medications that are known clinical organic anion-transporting polypeptide B1 (OATP1B1) and/or OATP1B3 inhibitors, concurrently or within 14 days of C1D1 of study drug(s).
17. Receipt of live attenuated vaccine (eg, tuberculosis Bacillus Calmette-Guerin vaccine, oral polio vaccine, measles, rotavirus, yellow fever) within 28 days of C1D1 of study drug(s).
18. Recipients of allogeneic or autologous stem cell transplantation or organ transplantation.

    For Part 2 SCCHN only:
19. Has progressive disease within 6 months of completion of curatively intended systemic treatment for locoregionally advanced SCCHN.
20. Has a life expectancy of less than 3 months and/or has rapidly progressive disease (eg, tumor bleeding, uncontrolled tumor pain) in the opinion of the treating investigator.
21. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) agent.
22. Participants with known dihydropyrimidine dehydrogenase (DPD) deficiency or thymidine phosphorylase gene (TYMP) mutations (Part 2B only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) and Based on TEAEs Severity | Up to approximately 68 months
  A severity grade is defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0. Grade 1 scales as Mild (asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2 scales as Moderate (minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living [ADL]); Grade 3 scales as Severe (severe or medically significant but not immediately life threatening hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 scales as Life-threatening consequences, urgent intervention indicated, and Grade 5 scales as Death related to Adverse Event (AE).
Number of Participants with Dose-Limiting Toxicities (DLTs) | Up to approximately 68 months
  A DLT will be defined as any of the TEAEs, but not limited to, those that occur during Cycle 1 and are considered by the investigator to be at least possibly related to dazostinag as a SA or in combination with pembrolizumab. TEAEs meeting DLT definitions occurring in Cycle 2 or later will be considered in the determination of the RDE of dazostinag, both in the dazostinag SA and the combination with pembrolizumab arms. Toxicity will be evaluated according to NCI CTCAE version 5.0.
Number of Participants Reporting One or More Treatment Emergent Serious Adverse Event (SAEs) | Up to approximately 68 months
Number of Participants With one or More TEAEs Leading to Dose Modifications and Treatment Discontinuations | Up to approximately 68 months

SECONDARY OUTCOMES:
Dose Escalation, Japan Safety Lead-in, and Expansion Phases: Overall Response Rate (ORR) | Up to approximately 68 months
  ORR is defined as the percentage of participants who achieve confirmed complete response (cCR) + confirmed partial response (cPR) during the study in response-evaluable population. ORR will be assessed based on Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1.
Dose Escalation, Japan Safety Lead-in, and Expansion Phases: Disease Control Rate (DCR) | Up to approximately 68 months
  DCR is defined as the percentage of participants who achieve cCR + cPR + stable disease (SD) greater than (>) 6 weeks during the study in response-evaluable population. The DCR will be assessed based on RECIST version 1.1.
Dose Escalation, Japan Safety Lead-in, and Expansion Phases: Duration of Response (DOR) | Up to approximately 68 months
  DOR is the time from the date of first documentation of a cPR or better to the date of first documentation of progressive disease for responders (cPR or better). Responders without documentation of progressive disease will be censored at the date of last response assessment that is SD or better. DOR will be assessed based on RECIST version 1.1.
Dose Escalation, Japan Safety Lead-in, and Expansion Phases: Time to Response (TTR) | Up to approximately 68 months
  TTR is defined as the time from the date of first dose administration to the date of first documented cPR or better by the investigator. TTR will be assessed based on RECIST version 1.1.
Expansion Phase Only: Progression-Free Survival (PFS) | Up to approximately 29 months
  PFS is defined as the time from the date of first dose administration to the date of first documented disease progression or death due to any cause, whichever occurs first.
Expansion Phase Only: Overall Survival (OS) | Up to approximately 29 months
  OS is defined as the time from the date of first dose administration to the date of death.
Expansion Phase Only: OS Rate at 12 Months | Up to 29 months
  12-month OS rate is defined as the percentage of participants who are still alive at 12 months from their first dose administration.
Expansion Phase Only: OS Rate at 6 Months | Up to 29 months
  6-month OS rate is defined as the percentage of participants who are still alive at 6 months from their first dose administration.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (61):
- United States (25):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - UCI Health - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center, Santa Monica, California
  - SCRI - HealthOne Denver, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Cancer Institute at Memorial Hospital West - Cancer Institute/Radiology Oncology, Gainesville, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Maryland Marlene and Stewart Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute - Lawrence and Idell Weisberg Cancer Treatment Center, Detroit, Michigan
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - University of Cincinnati Health Barrett Cancer Center, Cincinnati, Ohio
  - West Chester Hospital, West Chester, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Virginia Cancer Specialists, P.C. - Fairfax, Fairfax, Virginia
- Klinikum Wels-Grieskirchen, Wels, Upper Austria, Austria
- Canada (3):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Sheng
  - Sixth Affiliated Hospital of Sun Yat-Sen University/Guangdong Gastrointestinal Hospital, Guangzhou, Guangzhou Sheng
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - West China School of Medicine - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- France (10):
  - Centre Hospitalier Regional et Universitaire de Besancon - Hopital Jean-Minjoz, Besançon
  - Hopital Saint-Andre, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Centre de Lutte contre le Cancer - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital de la Timone, Marseille
  - Hopital Saint-Antoine, Paris
  - Institut de Cancerologie de lOuest - Saint-Herblain - Site Rene Gauducheau, Saint-Herblain
  - Gustave Roussy, Villejuif
  - Hopital Foch, Suresnes, Île-de-France Region
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- National Cancer Center Hospital, Chuo-Ku, Tokyo, Japan
- Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship, Poland
- PanOncology Trials: Universidad de Puerto Rico - Centro Comprensivo de Cancer, San Juan, Puerto Rico
- Switzerland (4):
  - Kantonsspital Sankt Gallen, Sankt Gallen, Canton of St. Gallen
  - Inselspital Universitatsspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne
- United Kingdom (4):
  - Queen's University Belfast, Belfast, Northern Ireland
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University College London Hospitals NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Carideo Cunniff E, Sato Y, Mai D, Appleman VA, Iwasaki S, Kolev V, Matsuda A, Shi J, Mochizuki M, Yoshikawa M, Huang J, Shen L, Haridas S, Shinde V, Gemski C, Roberts ER, Ghasemi O, Bazzazi H, Menon S, Traore T, Shi P, Thelen TD, Conlon J, Abu-Yousif AO, Arendt C, Shaw MH, Okaniwa M. TAK-676: A Novel Stimulator of Interferon Genes (STING) Agonist Promoting Durable IFN-dependent Antitumor Immunity in Preclinical Studies. Cancer Res Commun. 2022 Jun 23;2(6):489-502. doi: 10.1158/2767-9764.CRC-21-0161. eCollection 2022 Jun. PMID 36923556
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603d4db2bf003ab4a3a7